CLINICAL TRIAL: NCT06729515
Title: Rhomboid Intercostal Block with Subserratus Plane Block in Bariatric Surgery: a Three-arm Prospective Randomized Comparative Study
Brief Title: Rhomboid Intercostal Block with Subserratus Plane Block in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Head of Research, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-MER-116
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity/therapy
Keywords: patient-controlled analgesia; continuous epidural analgesia; the rhomboid intercostal block combined with subserratus plane block; bariatric surgery; numerical rating scale
MeSH Terms: conditions — Obesity | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Intervention Model Description: PCA group Immediately post-surgery, patients in the PCA group received a programmed PCA infusion (YG-B-3; Jiangsu Yaguang Medical Device Co., Ltd., China) containing either ketorolac (180 mg) or sufentanil (200 µg) in 100 mL, delivered as a 2 mL/h basal infusion with 0.5 mL boluses; lockout interval: 15 min.
  CEA group Following epidural catheter placement in the operating room, the CEA group received an initial bolus of 2% lidocaine (3 mL). Once sensory blockade was confirmed, continuous epidural infusion of 0.1% ropivacaine (8 mL/h) commenced.
  RISS group RISS blocks were performed at the T4-T10 level under ultrasound guidance (EPIQ5 with L12-4 linear 7.5 MHz transducer; Philips Healthcare, Best, Netherlands). A 19-gauge, 40-cm catheter was advanced 3-5 cm beyond the needle tip into the subserratus plane, its position confirmed by injecting 5 mL of 0.2% ropivacaine. A further 15 mL of 0.2% ropivacaine was then administered. The catheter was connected to a PCA pump programmed to deliver
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PCA group (Active Comparator): patient-controlled analgesia
  Interventions: Device: PCA
- CEA group (Active Comparator): continuous epidural analgesia
  Interventions: Device: CEA
- RISS group (Experimental): the rhomboid intercostal block combined with subserratus plane block
  Interventions: Device: RISS

INTERVENTIONS:
Device: PCA — Immediately post-surgery, patients in the PCA group received a programmed PCA infusion (YG-B-3; Jiangsu Yaguang Medical Device Co., Ltd., China) containing either ketorolac (180 mg) or sufentanil (200 µg) in 100 mL, delivered as a 2 mL/h basal infusion with 0.5 mL boluses; lockout interval: 15 min.
  Arms: PCA group
Device: CEA — Following epidural catheter placement in the operating room, the CEA group received an initial bolus of 2% lidocaine (3 mL). Once sensory blockade was confirmed, continuous epidural infusion of 0.1% ropivacaine (8 mL/h) commenced.
  Arms: CEA group
Device: RISS — RISS blocks were performed at the T4-T10 level under ultrasound guidance (EPIQ5 with L12-4 linear 7.5 MHz transducer; Philips Healthcare, Best, Netherlands). A 19-gauge, 40-cm catheter was advanced 3-5 cm beyond the needle tip into the subserratus plane, its position confirmed by injecting 5 mL of 0.2% ropivacaine. A further 15 mL of 0.2% ropivacaine was then administered. The catheter was connected to a PCA pump programmed to deliver a 7 mL/h basal infusion with 2 mL boluses; lockout interval: 30 min.
  Arms: RISS group

SUMMARY:
Standard analgesic techniques such as patient-controlled analgesia (PCA) and continuous epidural analgesia (CEA) are effective but associated with considerable side effects, including nausea, hypotension, and respiratory depression. This study aimed to evaluate the efficacy and safety of the rhomboid intercostal block combined with subserratus plane block (RISS) compared to PCA and CEA for postoperative analgesia in bariatric surgery.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, non-inferiority and superiority trial compared PCA, CEA, and RISS blocks for postoperative analgesia in bariatric surgery patients recruited at Baogang Hospital, Inner Mongolia. The study, approved by the Baogang Hospital Medical Ethics Committee (2022-MER-116; October 16, 2022), adhered to the Declaration of Helsinki and CONSORT guidelines. All participants provided informed consent.

This study included 144 patients (January-December 2023) undergoing elective bariatric surgery at Baogang Hospital, Inner Mongolia.

Patients were randomly assigned (1:1:1) to one of three groups: (1) PCA, (2) CEA, and (3) RISS block. Randomization was performed using a sequentially numbered, concealed allocation sequence generated from a random number table.

General anesthesia was induced with propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 µg/kg i.v.), followed by endotracheal intubation. Anesthesia was maintained with sevoflurane or desflurane, titrated to maintain a bispectral index (BIS) target. Remifentanil (0.05-0.2 µg/kg/min) was infused to maintain mean arterial pressure and heart rate within ±20% of baseline values. Mechanical ventilation was initiated using pressure-regulated volume control (PRVC) mode (Aestiva; GE Healthcare, Waukesha, WI, USA) with tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H₂O, inspiratory-expiratory ratio 1:2, respiratory rate 16 breaths per minute, and inspired oxygen fraction 0.41. The patient was positioned in a reverse Trendelenburg position (20-25° head-up tilt) and pneumoperitoneum was established with carbon dioxide at 10-15 mmHg.

PCA group Immediately post-surgery, patients in the PCA group received a programmed PCA infusion (YG-B-3; Jiangsu Yaguang Medical Device Co., Ltd., China) containing either ketorolac (180 mg) or sufentanil (200 µg) in 100 mL, delivered as a 2 mL/h basal infusion with 0.5 mL boluses; lockout interval: 15 min.

CEA group Following epidural catheter placement in the operating room, the CEA group received an initial bolus of 2% lidocaine (3 mL). Once sensory blockade was confirmed, continuous epidural infusion of 0.1% ropivacaine (8 mL/h) commenced.

RISS group RISS blocks were performed at the T4-T10 level under ultrasound guidance (EPIQ5 with L12-4 linear 7.5 MHz transducer; Philips Healthcare, Best, Netherlands). A 19-gauge, 40-cm catheter was advanced 3-5 cm beyond the needle tip into the subserratus plane, its position confirmed by injecting 5 mL of 0.2% ropivacaine. A further 15 mL of 0.2% ropivacaine was then administered. The catheter was connected to a PCA pump programmed to deliver a 7 mL/h basal infusion with 2 mL boluses; lockout interval: 30 min.

In the postanesthesia care unit (PACU), arterial blood pressure, heart rate, and the incidence of postoperative nausea and vomiting (PONV) were monitored and recorded. Symptomatic treatment was administered for hypotension, bradycardia, and PONV as needed.

Primary outcomes were rest and dynamic pain scores (numerical rating scale [NRS] ) at 4, 8, 12, and 24 hours postoperatively. Secondary outcomes included cumulative morphine equivalent dose (mg i.v.) at 4, 8, 12, and 24 hours postoperatively; incidence of postoperative nausea and vomiting (PONV); ondansetron use (mg); and quality of sleep on the first postoperative night (Likert scale, 1-5). Superiority and non-inferiority analyses were performed for all outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-41 years
* ASA I-III
* body mass index (BMI) ≥27.5 kg/m² or BMI <27.5 kg/m² with obesity-related comorbidities (type 2 diabetes mellitus, hypertension, obstructive sleep apnea, or non-alcoholic fatty liver disease)
* failure to achieve significant weight loss with conservative management (diet and/or pharmacotherapy)
* the capacity for postoperative care and lifestyle modification

Exclusion Criteria:

* severe cardiopulmonary or hepatic disease
* untreated major psychiatric disorders or active substance abuse potentially affecting postoperative lifestyle management; pregnancy or intention to conceive
* inability to complete long-term follow-up or lifestyle adjustments; or inability to obtain complete trial data
* Patients who refused to provide written informed consent were excluded

Ages: 20 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
NRS | Postoperative 4th hour, postoperative 8th hour, postoperative 12th hour, postoperative 24th hour
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Likert scale | Postoperative 4th hour, postoperative 8th hour, postoperative 12th hour, postoperative 24th hour
  quality of sleep on the first postoperative night (Likert scale, 1-5). Likert scale where 1=very dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied and 5=very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: January 2025-January 2026
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.

REFERENCES:
- Available data/document: Individual Participant Data Set — https://figshare.com/s/46ea85c406ec97afc17a